CLINICAL TRIAL: NCT04870489
Title: Fractional Ablative CO2 Laser Treatment for Acne Scars in Patients Receiving Oral Isotretinoin
Brief Title: Combined Treatment With CO2 Laser and Isotretinoin for Acne Scars
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0629-17
Record Dates: First submitted 2021-04-12; First posted 2021-05-03 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-04

CONDITIONS: Acne Vulgaris
Keywords: acne vulgaris;scars; CO2 laser; ISOTRETINOIN;treatments
MeSH Terms: conditions — Acne Vulgaris | interventions — Isotretinoin; Lasers, Gas

STUDY DESIGN:
Intervention Model Description: Patients are treated with Isotretinoin for at least 2 months prior to starting Co2 laser treatment, then they receive laser treatment on one side of the face (randomized) while still taking Isotretinoin; 6 months after cessation of Isotretinoin or any other treatment they are then treated with Co2 laser only on the second side of the face
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Isotretinoin + Co2 ablative laser (Active Comparator): Isotretinoin treatment while being treated with CO2 laser
  Interventions: Combination Product: Isotretinoin and CO2 laser
- Co2 ablative laser (Active Comparator): 6 months to 1 year without isotretinoin treatments to start second side of face with CO2 ablative laser only
  Interventions: Device: Co2 laser

INTERVENTIONS:
Combination Product: Isotretinoin and CO2 laser — Patients must complete at least 2 months of Isotretinoin prior to starting the study and then continue it for the duration of the 3 months of treatment with the CO2 laser.
  Arms: Isotretinoin + Co2 ablative laser
Device: Co2 laser — After 6-12 months of no treatment for acne the patient comes to do second side of face only laser treatment
  Arms: Co2 ablative laser

SUMMARY:
Isotretinoin is an FDA-approved vitamin A metabolite for the treatment of severe acne; acne that does not respond to other treatments and has a tendency to cause scarring.

Ablative laser treatment is another effective treatment against acne scarring. We believe that the combination of CO2 ablative laser treatment with oral isotretinoin for the treatment of scarring is not only safer but also more effective and leads to much more successful cosmetic results.

DETAILED DESCRIPTION:
Patients treated with Isotretinoin for at least 2 months with doses ranging from 20 mg-40 mg per day were treated with Co2 ablative laser on one side of the face (randomized). Patients will be treated with a single session using the fractional AcuPulse CO2 laser (AcuPulse; Lumenis Inc., Santa Clara, CA), with the AcuScan120™ scanner hand-piece and the Deep FX mode. The treatment areas will be cleansed with a mild cleanser and 70% alcohol. Local anesthesia, comprising a topical eutectic mixture of 2.5% lidocaine hydrochloric acid and 2.5% prilocaine cream (EMLA Cream; Astra Zeneca AB, Sweden), will be applied to the treated side of the face under occlusion before laser therapy. After an hour of application, the anesthetic cream will gently be removed, and then, to obtain a completely dry skin surface.Treatment parameters will be a flounce of 15 mj and density of 15% in single-pass treatment without overlapping pulse. Immediately after the treatment, gauzes moistened with cold saline solution must be gently applied (without rubbing) on the skin for 15-20 minutes. Thereafter a thin layer of mupirocin 2% ointment (TEVA PHARMACEUTICAL INDUSTRIES LTD, ISRAEL) will be applied on the skin.

After the procedure, a visual analog scale (VAS) will be used to determine the amount of pain felt by the participants. No pain will be scored as 0, and intolerable pain will be scored as 10 in this scale. Photographs will be taken at baseline; before each treatment; and 6 months after the last treatment. Acne scars will be graded by using the Quantitative Global Acne Scarring Grading System, which takes into account the quantity and type of scar based on a point system (13). With this grading scale, the total score can vary from 0 to 84. The overall score will be determined as the "acne scar score". All assessments will be done by two independent physicians and the mean value of the two assessments will be calculated. A 25% or less decrease in the acne scar score was defined as "mild improvement", 26-50% decrease as "moderate improvement", 51-75% decrease as "significant improvement", and over 75% as "near total improvement". Lack of decrease in the acne scar score was defined as "no change" and an increase in the score was defined as "worsening".

Subjective self-assessment by the participants were done 6 months after the last treatment and was scored as follows: - 1 as "worsening", 0 as "no change", 1 as "mild improvement", 2 as "moderate improvement", 3 as "significant improvement ", and 4 as "near total improvement". At this point, all patients will be 6 months after cessation of oral isotretinoin and will be treated with CO2 laser to the second half of the face with the same treatment parameters All patients will receive CO2 laser treatment once a month for 3 consecutive months (LASER treatment will be identical to the treatment mentioned above for the first half of the face).

The LASER treatment for the second half of the face will be also evaluated by two independent physicians and will be compared to the first side of the face which was previously treated. Both physicians will not be aware as to which side of the face is treated with laser during oral intake of isotretinoin and which side is not.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Age 15-60 years old
* Male/Female
* Acne moderate to severe with scarring
* Finished at least 2 months of treatment with Isotretinoin

Exclusion Criteria:

* Prior laser treatment for acne scarring
* Patients that have a tendency to have abnormal scarring
* Patients that are immunosuppressed or patients receiving immunosuppressive treatment
* Prior radiotherapy treatment to affected area
* Infected acne
* Rosacea

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative Global Acne Scarring Grading System | Photographs taken at baseline; before each treatment; and 6 months after the last treatment
  With this acne scars grading scale, the total score can vary from 0 to 84. The overall score will be determined as the "acne scar score". A 25% or less decrease in the acne scar score was defined as "mild improvement", 26-50% decrease as "moderate improvement", 51-75% decrease as "significant improvement", and over 75% as "near total improvement"

CONTACTS AND LOCATIONS:
Overall Officials: Eli Sprecher, Professor, Study Chair — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv sourasky medical center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
sex, age, acne severity, acne disease duration, accumulated isotretinoin dose prior to co2 laser and at the end of treatment, VAS score, skin type, weight, medical history

REFERENCES:
- [Background] Waldman A, Bolotin D, Arndt KA, Dover JS, Geronemus RG, Chapas A, Iyengar S, Kilmer SL, Krakowski AC, Lawrence N, Prather HB, Rohrer TE, Schlosser BJ, Kim JYS, Shumaker PR, Spring LK, Alam M. ASDS Guidelines Task Force: Consensus Recommendations Regarding the Safety of Lasers, Dermabrasion, Chemical Peels, Energy Devices, and Skin Surgery During and After Isotretinoin Use. Dermatol Surg. 2017 Oct;43(10):1249-1262. doi: 10.1097/DSS.0000000000001166. PMID 28498204
- [Background] Fife D. Practical evaluation and management of atrophic acne scars: tips for the general dermatologist. J Clin Aesthet Dermatol. 2011 Aug;4(8):50-7. PMID 21909457
- [Background] Tasoula E, Gregoriou S, Chalikias J, Lazarou D, Danopoulou I, Katsambas A, Rigopoulos D. The impact of acne vulgaris on quality of life and psychic health in young adolescents in Greece. Results of a population survey. An Bras Dermatol. 2012 Nov-Dec;87(6):862-9. doi: 10.1590/s0365-05962012000600007. PMID 23197205
- [Background] Strauss JS, Krowchuk DP, Leyden JJ, Lucky AW, Shalita AR, Siegfried EC, Thiboutot DM, Van Voorhees AS, Beutner KA, Sieck CK, Bhushan R; American Academy of Dermatology/American Academy of Dermatology Association. Guidelines of care for acne vulgaris management. J Am Acad Dermatol. 2007 Apr;56(4):651-63. doi: 10.1016/j.jaad.2006.08.048. Epub 2007 Feb 5. PMID 17276540
- [Background] Amichai B, Shemer A, Grunwald MH. Low-dose isotretinoin in the treatment of acne vulgaris. J Am Acad Dermatol. 2006 Apr;54(4):644-6. doi: 10.1016/j.jaad.2005.11.1061. PMID 16546586
- [Background] Goldstein JA, Socha-Szott A, Thomsen RJ, Pochi PE, Shalita AR, Strauss JS. Comparative effect of isotretinoin and etretinate on acne and sebaceous gland secretion. J Am Acad Dermatol. 1982 Apr;6(4 Pt 2 Suppl):760-5. doi: 10.1016/s0190-9622(82)70066-0. PMID 6461679
- [Background] Jones DH, King K, Miller AJ, Cunliffe WJ. A dose-response study of I3-cis-retinoic acid in acne vulgaris. Br J Dermatol. 1983 Mar;108(3):333-43. doi: 10.1111/j.1365-2133.1983.tb03973.x. PMID 6219690
- [Background] Layton AM, Knaggs H, Taylor J, Cunliffe WJ. Isotretinoin for acne vulgaris--10 years later: a safe and successful treatment. Br J Dermatol. 1993 Sep;129(3):292-6. doi: 10.1111/j.1365-2133.1993.tb11849.x. PMID 8286227
- [Background] Abergel RP, Meeker CA, Oikarinen H, Oikarinen AI, Uitto J. Retinoid modulation of connective tissue metabolism in keloid fibroblast cultures. Arch Dermatol. 1985 May;121(5):632-5. PMID 3994409
- [Background] Cruz NI, Korchin L. Inhibition of human keloid fibroblast growth by isotretinoin and triamcinolone acetonide in vitro. Ann Plast Surg. 1994 Oct;33(4):401-5. doi: 10.1097/00000637-199410000-00007. PMID 7810956
- [Background] Sporn MB, Roberts AB, Roche NS, Kagechika H, Shudo K. Mechanism of action of retinoids. J Am Acad Dermatol. 1986 Oct;15(4 Pt 2):756-64. doi: 10.1016/s0190-9622(86)70231-4. PMID 3021829
- [Background] Manstein D, Herron GS, Sink RK, Tanner H, Anderson RR. Fractional photothermolysis: a new concept for cutaneous remodeling using microscopic patterns of thermal injury. Lasers Surg Med. 2004;34(5):426-38. doi: 10.1002/lsm.20048. PMID 15216537
- [Background] Chandrashekar BS, Varsha DV, Vasanth V, Jagadish P, Madura C, Rajashekar ML. Safety of performing invasive acne scar treatment and laser hair removal in patients on oral isotretinoin: a retrospective study of 110 patients. Int J Dermatol. 2014 Oct;53(10):1281-5. doi: 10.1111/ijd.12544. Epub 2014 Jul 11. PMID 25039864
- [Result] Layton AM, Henderson CA, Cunliffe WJ. A clinical evaluation of acne scarring and its incidence. Clin Exp Dermatol. 1994 Jul;19(4):303-8. doi: 10.1111/j.1365-2230.1994.tb01200.x. PMID 7955470